CLINICAL TRIAL: NCT07317375
Title: Effectiveness of Stanley Paris Manual Therapy Concept Versus Conventional Physiotherapy in Pain Reduction and Functional Improvement in Grade II Knee Osteoarthritis
Brief Title: Effectiveness of Stanley Paris Manual Therapy vs. Conventional Physiotherapy in Reducing Pain and Improving Function in Grade II Knee Osteoarthritis
Acronym: SPMT vs CPT in
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibadat International University, Islamabad (Other)
Collaborators: Helping Hand Institute of Rehabilitation Sciences (Other)
Responsible Party: Principal Investigator, Dr Abdul Haseeb Bhutta, ASSISTANT PROFESSOR / HOD PHYSICAL THERAPY DEPARTMENT, Ibadat International University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIUI/RERC/ADT/2025/07/178-1
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; knee; Stanley Paris
MeSH Terms: conditions — Osteoarthritis | interventions — Musculoskeletal Manipulations; Transcutaneous Electric Nerve Stimulation; High-Energy Shock Waves; Pliability; Exercise

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with a parallel-group design involving 50 participants diagnosed with Grade II Knee Osteoarthritis. Participants will be randomly assigned into two groups: Group A will receive the Stanley Paris Manual Therapy Concept, and Group B will receive Conventional Physiotherapy. Both groups will undergo supervised sessions 2-3 times per week for 6-8 weeks. Randomization will be computer-generated, and outcome assessors will be blinded to group allocation. The study follows a prospective, single-blinded, two-arm model, comparing manual therapy-based rehabilitation with traditional physiotherapy for pain reduction, functional improvement, and enhanced quality of life in knee osteoarthritis patients.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will use a quadruple-blind design in which the participants, care providers, investigators, and outcomes assessors will all be masked to group allocation. Randomization will be conducted using a coded allocation system managed by an independent coordinator. Intervention protocols will be standardized and labeled by code to ensure blinding of treatment identity. Data collection and analysis will be performed without revealing group assignments to maintain objectivity and reduce bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stanley Paris group (Experimental): Participants in this group will receive treatment based on the Stanley Paris Manual Therapy Concept, which emphasizes hands-on techniques to restore joint biomechanics and improve movement patterns. Interventions will include joint mobilization (Maitland and Kaltenborn grades II-IV), soft tissue and myofascial release, neural mobilization, proprioceptive training, and functional movement retraining. Sessions will be conducted 4 times per week for 6 weeks by trained physiotherapists following a standardized treatment protocol.
  Interventions: Other: Hands-on manual therapy including joint mobilization, soft tissue and neural mobilization, and movement retraining based on the Stanley Paris Concept.
- Conventional Physical Therapy (Active Comparator): Participants in this group will receive Conventional Physiotherapy, including electrotherapy modalities (TENS, ultrasound, heat/cold therapy), general strengthening exercises, range-of-motion and flexibility exercises, and basic balance training. The focus will be on pain reduction, muscle strengthening, and functional mobility improvement. Sessions will also be conducted 4 times per week for 6 weeks following standard clinical practice guidelines for knee osteoarthritis management.
  Interventions: Other: Conventional Physiotherapy Standard physiotherapy care including electrotherapy modalities (TENS, ultrasound), strengthening, flexibility, and balance training exercises.

INTERVENTIONS:
Other: Hands-on manual therapy including joint mobilization, soft tissue and neural mobilization, and movement retraining based on the Stanley Paris Concept. — This intervention follows the Stanley Paris Manual Therapy Concept, a hands-on approach emphasizing biomechanical correction and functional movement restoration. Treatment will include Maitland and Kaltenborn joint mobilization (Grades II-IV), patellar glides, soft tissue and myofascial release, neural mobilization, and movement pattern retraining. Sessions will also include proprioceptive and balance exercises, functional strengthening, and patient education on posture and joint protection. Each participant will receive 4 sessions per week for 6 weeks, lasting approximately 45-60 minutes each, delivered by trained manual therapists using a standardized protocol.
  Other Names: Manual Therapy; Stanley Paris Approach; joint Mobilization and Movement Re-education
  Arms: Stanley Paris group
Other: Conventional Physiotherapy Standard physiotherapy care including electrotherapy modalities (TENS, ultrasound), strengthening, flexibility, and balance training exercises. — This intervention consists of standard physiotherapy treatment commonly used for Grade II Knee Osteoarthritis. It includes electrotherapy modalities such as TENS, ultrasound, and hot/cold therapy, along with therapeutic exercises for strengthening, flexibility, and balance. Exercises include open-chain and closed-chain strengthening, range-of-motion activities, and static stretching. Participants will receive 4 supervised sessions per week for 6 weeks, each lasting 45-60 minutes, administered by qualified physiotherapists following evidence-based clinical practice guidelines.
  Other Names: Routine Physiotherapy; Standard Physical Therapy; Exercise and Electrotherapy Program
  Arms: Conventional Physical Therapy

SUMMARY:
This study aims to compare two different physiotherapy approaches for people suffering from Grade II Knee Osteoarthritis (OA) - a condition that causes knee pain, stiffness, and difficulty in walking.

The first approach is the Stanley Paris Manual Therapy Concept, which involves hands-on treatment techniques such as joint mobilization, soft tissue massage, and movement correction. The second is Conventional Physiotherapy, which uses traditional exercises and electrotherapy (like heat, ultrasound, or TENS) to reduce pain and improve strength.

The study will include 50 patients aged 40-60 years who have moderate knee osteoarthritis. They will be randomly divided into two groups - one receiving manual therapy and the other receiving conventional physiotherapy - for 6 to 8 weeks.

Researchers will measure pain, knee function, range of motion, balance, and quality of life before and after treatment to see which method gives better results.

By identifying which therapy works more effectively, this study will help patients, families, and healthcare providers choose the most beneficial and evidence-based treatment for improving movement, reducing pain, and enhancing daily living activities in people with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a common degenerative joint disorder that causes pain, stiffness, and loss of mobility, often leading to functional limitations and reduced quality of life. In Grade II OA, cartilage damage is moderate and potentially reversible through appropriate rehabilitation strategies. This stage offers an important opportunity for physiotherapy interventions to restore function and delay further joint deterioration.

The Stanley Paris Manual Therapy Concept emphasizes a biomechanical and hands-on approach to rehabilitation. It includes joint mobilization, soft tissue manipulation, neural mobilization, and correction of faulty movement patterns to restore normal joint motion and neuromuscular control. In contrast, Conventional Physiotherapy typically focuses on pain management using electrotherapy modalities, strengthening exercises, and general mobility training.

This randomized controlled trial (RCT) is designed to compare the effectiveness of these two treatment approaches in individuals with Grade II knee osteoarthritis. Fifty participants will be randomly allocated into two equal groups: one receiving the Stanley Paris manual therapy and the other receiving conventional physiotherapy, for a period of 6-8 weeks. Standardized assessment tools - including the Visual Analog Scale (VAS) for pain, the Knee Injury and Osteoarthritis Outcome Score (KOOS) for function and quality of life, and the Berg Balance Scale for proprioception and stability - will be used to evaluate outcomes at baseline, mid-intervention, and post-intervention.

The study will generate clinical evidence on whether manual therapy provides superior outcomes in terms of pain relief, functional improvement, and patient satisfaction compared to conventional physiotherapy. Results are expected to assist clinicians in developing more effective rehabilitation protocols for managing knee osteoarthritis and improving patients' independence and overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Grade II knee osteoarthritis based on radiographic and clinical criteria.
* Participants experiencing knee pain for at least three months.
* Ability to walk independently without assistive devices.
* Willingness to participate in a structured physiotherapy program.

Exclusion Criteria:

* Presence of Grade III or IV knee osteoarthritis.
* History of knee surgery or joint replacement.
* Rheumatoid arthritis or other inflammatory joint diseases.
* Neurological conditions affecting lower limb function.
* Contraindications to manual therapy or exercise interventions.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction Measured by Visual Analog Scale (VAS) | Change in pain intensity from baseline to 4th week and 8 weeks
  The Visual Analog Scale (VAS) will be used to assess the intensity of knee pain. Participants will mark their pain level on a 10 cm line ranging from 0 ("no pain") to 10 ("worst imaginable pain"). Pain scores will be recorded at baseline, after 4 weeks, after 8 weeks of treatment.
Functional Improvement Measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change in KOOS scores from baseline to 4th weeks and 8 weeks.
  The KOOS questionnaire will assess knee function, daily living activities, sports and recreation function, and knee-related quality of life. Each subscale is scored from 0 (extreme problems) to 100 (no problems).
Knee Range of Motion Measured by Goniometer | Change from baseline to 4th weeks and 8 weeks post-intervention.
  Active knee flexion and extension will be measured using a standard universal goniometer to assess joint mobility.
Balance and Proprioception Measured by Berg Balance Scale | Change from baseline to 4th week and 8 weeks post-intervention.
  The Berg Balance Scale (14 items, score range 0-56) will assess participants' static and dynamic balance. Higher scores indicate better balance and lower fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad Nazim Farooq, Ph.D., Study Director — Ibadat International University, Islamabad
Locations (1):
- Ibadat international University islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the results of this study - including demographic data, baseline characteristics, intervention details, and outcome measures (VAS, KOOS, Range of Motion, and Berg Balance Scale scores) - may be shared. No personally identifiable information will be disclosed. Data will be available upon reasonable request from qualified researchers for academic or clinical research purposes following publication of the main study results.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: February 2026
Access Criteria: On demand IPD will be shared with journals editor